CLINICAL TRIAL: NCT04166292
Title: A Prospective, Monocentric, Uncontrolled Clinical Investigation to Evaluate the Efficacy and Safety of Stylage® XL Lidocaïne for the Restoration and/or Augmentation of Facial Volume
Brief Title: The Evaluation of Efficacy and Safety of Stylage® XL Lidocaïne for the Restoration and/or Augmentation of Facial Volume
Acronym: BeautyVolume
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoires Vivacy (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-A01404-53
Record Dates: First submitted 2019-11-14; First posted 2019-11-18 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Aging; Healthy
Keywords: augmentation; restoration; dermal filler; face; cheekbone; chin; mandibular angle; hyaluronic acid
MeSH Terms: conditions — Facies

STUDY DESIGN:
Masking Description: The facial volume loss will be retrospectively assessed by a blinded independent evaluator using the Facial Volume Loss Scale (FLVS) on 3D photographs from V1 (D0 before) and at the following visits: V2 (D30 before), V3 (D90), V4 (D180), V5 (D360) and V6 (D540). The evaluator is blinded to treatment and visit number.
  The overall improvement level will be retrospectively assessed by a blinded independent evaluator using the GAIS on 3D photographs at the following visits (in comparison with 3D photographs before injection): V2 (D30 before), V3 (D90), V4 (D180), V5 (D360) and V6 (D540). The evaluator is blinded to treatment and visit number.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treated face (Experimental): The device will be injected on V1 (D0) in the cheekbones (upper part of the cheek) for all subjects and in the chin for 20 subjects minimum and if needed (optional areas) in the temple, and facial oval (mandibular angle and border). A touch-up is possible in one or several of these areas on V2 (M1). Optional treated areas will be at the discretion of subjects and injectors.
  Interventions: Device: Stylage® XL Lidocaïne

INTERVENTIONS:
Device: Stylage® XL Lidocaïne — On V1 (D0), a total volume of 8 mL maximum can be used per subject on the whole face.
  On V2 (M1), a possible touch-up can be made according to the injector and subject's opinion which cannot exceed 4 ml.

SUMMARY:
Stylage® XL Lidocaïne is a CE-marketed hyaluronic acid gel indicated for the restoration or augmentation of facial volume by injection into the deep dermis or subcutaneously. Lidocaine hydrochloride is intended to reduce the pain associated with the injection.

In this study 40 healthy subjects between the age of 30 and 65 years, presenting a volume deficit on the face as evaluated by the investigator at inclusion in the study, who have given his/her informed consent and met all the eligibility criteria, will be enrolled.

Subjects will come to a total of 6 visits over a period of 18 months and a screening visit prior to baseline injection. The facial volume variation after baseline injection will be assessed. Treatment responders rate, Global Aesthetic Improvement, volume on the cheekbones, volume on the chin and chin angle (for applicable subjects), subject's satisfaction and safety will be also assessed.

DETAILED DESCRIPTION:
This is a prospective, uncontrolled, single site study with a blinded evaluator assessing the efficacy of Stylage® XL Lidocaïne on FVLS and GAIS clinical scoring.

The study duration by subject is 18 months with a screening visit (V0) before injection, the baseline visit (injection of Stylage® XL Lidocaïne, V1) and 5 follow-up visits after 1, 3, 6, 12 and 18 months (V2 to V6). At 1 month (V2) an optional touch-up may be done (if needed).

The primary endpoint is the facial volume variation from baseline (D0) to 6 months after treatment initiation measured by an independent evaluator on photographs using FVLS (Facial Volume Loss Scale).

Facial volume variation (evaluated by an independent evaluator) & treatment responder rate, Global Aesthetic Improvement (evaluated by the patient and the doctor), volume on the cheekbones and chin & chin angle (for applicable subjects), subject's satisfaction will be measured at all time-point with a FVLS, GAIS,3D QuantifiCare system, FACE-Q questionnaire (cheekbones and chin) respectively. Safety will be also assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Subject;
* Sex: male or female;
* Age: between 30 and 65 years;
* Subject having given freely and expressly his informed consent;
* Subject requiring injection on the cheekbones (upper part of the cheek);
* Subject with grade from 3 to 5 on the Facial Volume Loss Scale (FVLS);
* Subject, psychologically able to understand the study related information and to give a written informed consent;
* Subject affiliated to a health social security system;
* Female of childbearing potential should use a medically accepted contraceptive regimen since at least 12 weeks before the beginning of the study and during all the study;
* Subject agreeing to keep their usual cleansing / care products during the whole study period;
* Subject agreeing to apply a Sun Protection Factor (SPF) 50 cream during non-intensive exposure to sunlight.

Exclusion Criteria:

In terms of population

* Pregnant or nursing woman or planning a pregnancy during the study;
* Subject with a scar, moles or anything on the face which might interfere with the evaluation;
* Subject who had been deprived of their freedom by administrative or legal decision or who is under guardianship;
* Subject in a social or sanitary establishment;
* Subject participating to another research on human beings or who is in an exclusion period of one;
* Subject having received 4500 euros indemnities for participation in researches involving human beings in the 12 previous months, including participation in the present study.
* Intensive exposure to sunlight or Ultraviolet-rays (UV-rays) within the month before each visit;

In terms of associated pathology

* Subject suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study results;
* Subject with known history of or suffering from autoimmune disease and/or immune deficiency;
* Subject suffering from inflammatory and/or infectious cutaneous disorders in or near the studied zones (herpes, acne, mycosis, papilloma…). Subject with recurrent herpes is not eligible even if asymptomatic at time of inclusion;
* Subject prone to develop inflammatory skin conditions or having tendency to bleeding disorders
* Subject having history of allergy or anaphylactic shock including hypersensitivity to hyaluronic acid or to one of the components of the tested device;
* Subject having history of allergy or anaphylactic shock including hypersensitivity to amide-type local anaesthetics or antiseptic solution;
* Subject with a past history of streptococcal disease, such as acute rheumatic fever or recurrent sore throats;
* Subject with a tendency to develop keloids or hypertrophic scars;
* Subject with haemostatic disorder;
* Subject with porphyria;

Relating to previous or ongoing treatment

* Subject having received treatment with a laser, a dermabrasion, a surgery, a deep chemical peeling or other ablative procedure on the face within the past 12 months prior to inclusion;
* Subject having received injection with a resorbable filling product in the face area within the past 18 months prior to inclusion;
* Subject having received at any time injection with a slowly resorbable filling product (polylactic acid, calcium hydroxyapatite, combinations of hyaluronic acid (HA) and hypromellose, HA and dextran microbeads or HA and TriCalcium Phosphate (TCP), …) or with a non-resorbable filling product (polyacrylamide, silicone, combination of methacrylic polymers and collagen, polymer particles, …);
* Subject having received at any time a treatment with tensor threads on the face;
* Subject having started or changed her oral contraceptive or any other hormonal treatment during 12 weeks prior to inclusion;
* Subject under medications that reduce or inhibit hepatic metabolism;
* Subject under medications which may cause lipo-atrophy;
* Subject using medication such as aspirin, NSAIDs (ibuprofen, naproxen, …), antiplatelet agents, anticoagulants, vitamin C within one week prior to inclusion and agreeing not to take such treatments within 1 week prior to visit 2 (M1) or being a chronic user;
* Subject undergoing a topical treatment on the test area or a systemic treatment;

  * anti-histamines during the 2 weeks prior to study start;
  * immunosuppressors and/or corticoids during the 4 weeks prior to study start;
  * retinoids during the 6 months prior to study start.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-11-21 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2021-08-07 (Actual)

PRIMARY OUTCOMES:
Variation of facial volume | 6 months
  Facial volume variation from baseline to 6 months after treatment initiation measured by an independent evaluator on photographs using FVLS (Facial Volume Loss Scale). Graded scale from 1-5; 5 being the most severe

SECONDARY OUTCOMES:
Variation of facial volume | Month 1, Month 3, Month 12, Month 18
  Facial volume variation from baseline to 1, 3, 12 and 18 months after treatment initiation measured by an independent evaluator on photographs using FVLS scale.Graded scale from 1-5; 5 being the most severe
Treatment responders rate | Month 1, Month 3, Month 6, Month 12, Month 18
  Rate of treatment responders at 1, 3, 6, 12 and 18 months measured by an independent evaluator on photographs using FVLS scale. Graded scale from 1-5; 5 being the most severe
Global aesthetic improvement | Month 1, Month 3, Month 6, Month 12, Month 18
  Variation from baseline to 1, 3, 6, 12 and 18 months after treatment initiation of the global aesthetic improvement measured by an independent evaluator on photographs using the GAIS (Global Aesthetic Improvement Scale). 5 possibles grades : 1) Very much improved, 2) much improved, 3) improved, 4) no change, 5) worse
Patient self-assessed aesthetic improvement | Month 1, Month 3, Month 6, Month 12, Month 18
  Variation from baseline to 1, 3, 6, 12 and 18 months after treatment initiation of the global aesthetic improvement measured by subjects using the GAIS. 5 possibles grades : 1) Very much improved, 2) much improved, 3) improved, 4) no change, 5) worse
Variation of volume on the cheekbones, and on the chin for applicable subjects | Month 1, Month 3, Month 6, Month 12, Month 18
  Variation from baseline to 1, 3, 6, 12 and 18 months after treatment initiation of the volume on the cheekbones (upper part of the cheek) and on the chin, for applicable subjects, using the 3D QuantifiCare system.
Variation of the chin angle for applicable subjects | Month 1, Month 3, Month 6, Month 12, Month 18
  Variation from baseline to 1, 3, 6, 12 and 18 months after treatment initiation of the chin angle for applicable subjects using the 3D QuantifiCare system.
Evolution of subject's satisfaction | Month 1, Month 3, Month 6, Month 12, Month 18
  Evolution of subject's satisfaction from baseline to 1, 3, 6, 12 and 18 months after treatment initiation using the FACE-Q satisfaction with cheekbones and the FACE-Q satisfaction with chin questionnaires.
Report of adverse events | Month 1, Month 3, Month 6, Month 12, Month 18
  Evaluation of product tolerance by collection of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Alain-Ali MOJALLAL, MD, Principal Investigator
Locations (1):
- Laboratoire DERMSCAN, Villeurbanne, Rhône, France

IPD SHARING:
Plan to Share IPD: No